CLINICAL TRIAL: NCT07292974
Title: DYNAMIC CHANGES OF ENDOTHELIAL GLYCOCALYX AND INFLAMMATORY RESPONSE IN PATIENTS WITH ACUTE STROKE TREATED WITH MECHANICAL THROMBECTOMY
Brief Title: ENDOTHELIAL GLYCOCALYX AND INFLAMMATORY RESPONSE CHANGES IN PATIENTS WITH ACUTE STROKE UNDERGOING MECHANICAL THROMBECTOMY
Acronym: DEGIMT
Status: Not yet recruiting | Type: Observational
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: University Hospital Rijeka (Other); University of Rijeka (Other)
Responsible Party: Principal Investigator, Marijana Matas, MD, Clinical Hospital Centre Zagreb
Other Study IDs: uniri-iz-25-224
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Thrombectomy; Endothelial Glycocalyx
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute stroke patients: MT/ MT + thrombolysis/ thormbolysis only
  Interventions: Procedure: Mechanical thrombectomy

INTERVENTIONS:
Procedure: Mechanical thrombectomy — The concentrations of EG degradation products and inflammatory cytokines would be determined by the enzymatic immunoabsorption test method from peripheral blood and blood samples from cerebral circulation after reperfusion.

SUMMARY:
Ischemic stroke (IS) is one of the leading causes of mortality and disability. Treatment of IS is based on reperfusion methods, thrombolysis and mechanical thrombectomy (MT). However, there are significant limitations in their implementation and success. Also, there is a mismatch between successful recanalization of the blood vessel, recovery of the neurological status as well as treatment outcome. Precisely for these reasons, there is a need for a better understanding of pathophysiology events in the acute IS and for the development of new therapeutic procedures that would include neuroprotection, modification of the inflammatory response and preservation of the integrity of the blood-brain barrier. Acute IS occurs as a result of a blood vessel blockage, which leads to ischemic damage to the brain parenchyma. It causes an early inflammatory response that is extremely complex, involving a large number of inflammatory cytokines whose dynamics and role in the pathophysiology of IS are insufficiently investigated. It is known that inflammatory processes damage the endothelial glycocalyx (EG), a thin luminal layer of the endothelium that has numerous functions such as maintaining the integrity of blood vessels and regulating tone, and itself participates in the inflammatory response. In the brain, EG is a key regulator of the integrity of the blood-brain barrier, and its damage makes the barrier more permeable, which can lead to edema and the passage of potentially harmful substances. Clinical studies have shown that there is a possible relationship between the prognosis of patients with IS and the concentration of EG breakdown products in the peripheral blood. However, the relationship between changes in EG and the inflammatory process in the context of IS, and especially in relation to available treatment methods, remains unclear. The aim of the proposed study is to determine and analyze the dynamics of concentrations of EG degradation products and inflammatory cytokines in patients with acute IS during and after MT. This study would include all adult patients with acute IS who will undergo MT, and the concentrations of EG degradation products and inflammatory cytokines would be determined by the enzyme immunoassay method from peripheral blood and blood samples from the cerebral circulation after reperfusion. The obtained results will be correlated with the collected data on the neurological condition of the patient before and after the intervention, the type and course of the intervention performed, the course and duration of hospital treatment, the occurrence of complications and the outcome of treatment.

ELIGIBILITY:
Inclusion Criteria: all patients older than 18 years with a diagnosis of acute IS confirmed by brain CT or MRI, and to whom MT will be performed, regardless of whether they are previously received thrombolysis.

Exclusion Criteria: patients under the age of 18, patients with diagnosed with hemorrhagic stroke, patients with acute infection, autoimmune illness, malignant disease, trauma, pregnant women or patients who will refuse to participate in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients older than 18 years with a diagnosis of acute IS confirmed by brain CT or MRI, and to whom MT will be performed.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Concentrations of EG degradation products (syndecan 1, heparan sulfate) and the neovascularization factor VEGF in peripheral blood during the intervention and 24 hours after revascularization/attempted revascularization. | 24 hours
  To measure and analyze the concentrations of EG degradation products (syndecan 1, heparan sulfate) and the neovascularization factor VEGF in peripheral blood during the intervention and 24 hours after revascularization/attempted revascularization. Additionally, the concentrations of EG degradation products in a blood sample from the occlusion site after revascularization will be measured and analyzed.
Cytokine concentrations (IL 6, IL 10) | 24 hours
  Measure and analyze cytokine concentrations (IL 6, IL 10) in peripheral blood during the intervention and 24 hours after revascularization/attempted revascularization.

IPD SHARING:
Plan to Share IPD: No